CLINICAL TRIAL: NCT01455090
Title: Open-Label, Multiple-Dose, Dose Escalation Study to Evaluate the Pharmacodynamics, Pharmacokinetics, and Safety of Coadministration of BMS-650032, BMS-790052, and BMS-791325 When Administered for 24 or 12 Weeks in Treatment-Naïve Subjects Infected With Hepatitis C Virus Genotype 1
Brief Title: Study to Determine the Effectiveness and Safety of a Three Drug Antiviral Combination Therapy to Treat Hepatitis C Virus (HCV) Infected Patients Not Previously Treated With Currently Available Medications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI443-014; 2011-002788-11 (EudraCT Number)
Record Dates: First submitted 2011-10-18; First posted 2011-10-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — asunaprevir; daclatasvir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (13):
- Group 1:BMS-650032(200 mg)+BMS-790052(60 mg)+BMS-791325(75mg) (Experimental): BMS-650032 200 mg tablet by mouth twice daily for 24 Weeks
  BMS-790052 60 mg tablet by mouth once daily for 24 Weeks
  BMS 791325 75 mg table by mouth twice daily for 24 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 2:BMS-650032(200 mg)+BMS-790052(60 mg)+BMS-791325(75mg) (Experimental): BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 60 mg tablet by mouth once daily for 12 Weeks
  BMS 791325 75 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 3:BMS-650032(200 mg)+BMS-790052(60 mg)+BMS-791325(150mg) (Experimental): * Contingent upon review of safety data from all available treated subjects from Groups 1 and 2
  BMS-650032 200 mg tablet by mouth twice daily for 24 Weeks
  BMS-790052 60 mg tablet by mouth once daily for 24 Weeks
  BMS 791325 150 mg table by mouth twice daily for 24 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 4:BMS-650032(200 mg)+BMS-790052(60 mg)+BMS-791325(150mg) (Experimental): * Contingent upon review of safety data from all available treated subjects from Groups 1 and 2
  BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 60 mg tablet by mouth once daily for 12 Weeks
  BMS 791325 150 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 5:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(75mg) (Experimental): * Genotype 1 treatment-naive subjects
  BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 12 Weeks
  BMS 791325 75 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 6:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(150mg) (Experimental): * Genotype 1 treatment-naive subjects
  BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 12 Weeks
  BMS 791325 150 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 7:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(75mg) (Experimental): * Genotype 4 treatment-naive subjects
  BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 12 Weeks
  BMS 791325 75 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 8:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(150mg) (Experimental): * Genotype 4 treatment-naive subjects
  BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 12 Weeks
  BMS 791325 150 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group 9:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(75mg) (Experimental): * Genotype 1 treatment-null/non-responder subjects
  BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 12 Weeks
  BMS 791325 75 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group10:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(150mg) (Experimental): * Genotype 1 treatment-null/non-responder subjects
  BMS-650032 200 mg tablet by mouth twice daily for 12 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 12 Weeks
  BMS 791325 150 mg table by mouth twice daily for 12 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group11:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(75mg) (Experimental): * Genotype 1 treatment-null/non-responder subjects
  BMS-650032 200 mg tablet by mouth twice daily for 24 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 24 Weeks
  BMS 791325 75 mg table by mouth twice daily for 24 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Group12:BMS-650032(200 mg)+BMS-790052(30 mg)+BMS-791325(150mg) (Experimental): * Genotype 1 treatment-null/non-responder subjects
  BMS-650032 200 mg tablet by mouth twice daily for 24 Weeks
  BMS-790052 30 mg tablet by mouth twice daily for 24 Weeks
  BMS 791325 150 mg table by mouth twice daily for 24 Weeks
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325
- Grp13:BMS-650032(200mg)+BMS-790052(30mg)+BMS-791325(75mg)+RBV (Experimental): * Genotype 1 treatment-naive subjects
  BMS-650032 200 mg tablets orally twice daily 12 weeks
  BMS-790052 30 mg tablets orally twice daily 12 weeks
  BMS-791325 75 mg tablets orally twice daily 12 weeks
  Ribavirin (RBV) tablets orally weight based dosing daily 12 weeks [if subject is < 75 kg: 1000 mg per day orally (2 x 200 mg tablets in AM and 3 x 200 mg tablets in PM), or if ≥ 75 kg: 1200 mg per day orally (3 x 200 mg tablets in AM and 3 x 200 mg tablets in PM]
  Interventions: Drug: BMS-650032; Drug: BMS-790052; Drug: BMS-791325; Drug: Ribavirin

INTERVENTIONS:
Drug: BMS-650032
  Other Names: Asunaprevir (ASV)
Drug: BMS-790052
  Other Names: Daclatasvir (DCV)
Drug: BMS-791325
Drug: Ribavirin
  Other Names: Copegus®
  Arms: Grp13:BMS-650032(200mg)+BMS-790052(30mg)+BMS-791325(75mg)+RBV

SUMMARY:
The purpose of this study is to estimate the rate of sustained virologic response (SVR) SVR12, where SVR12 is defined as HCV RNA < LOQ (detectable or undetectable) 12 weeks post-treatment in Genotype 1 & Genotype 4 treatment naive patients, and Genotype (GT1) infected patients who are prior null responders to pegIFN/ribavirin

DETAILED DESCRIPTION:
IND numbers: 79,599; 101,943

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages ≥18 years of age
* Subjects who are naive to HCV treatment, defined as no previous exposure to an Interferon (IFN), Ribavirin (RBV); or any HCV-specific direct acting antiviral or experimental therapy or subjects who are null responders to previous pegylated Interferon alfa (pegIFNα) plus Ribavirin (RBV) treatment
* Subjects should have chronic hepatitis C (CHC) as documented by:

  1. Positive for anti-HCV antibody, HCV RNA, or a positive HCV genotype test at least 6 months prior to screening, and positive for HCV RNA and Anti-HCV antibody at the time of screening, or
  2. Positive for anti-HCV antibody and HCV RNA at the time of screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed prior to enrollment with evidence of CHC disease, such as the presence of fibrosis)
* HCV genotype 1a, 1b or 4 only
* HCV RNA viral load of ≥10,000 IU/mL at screening
* Have one of the following:

  1. Documented Fibrotest score of ≤0.72 and aspartate transferase (transminase) to platelet ratio index (APRI) ≤2; OR
  2. Documented liver biopsy within 36 months preceding Day 1 showing absence of cirrhosis OR
  3. Documented Fibroscan® ultrasound (where approved) within 12 months of screening showing absence of cirrhosis
* Body mass index (BMI) of 18.0 to 35.0 kg/m2, inclusive
* Subjects with compensated Child-Pugh A cirrhosis as documented by history of cirrhosis with any prior liver biopsy or Fibroscan® ultrasound (where approved) within 12 months prior to screening

Exclusion Criteria:

* Evidence of a medical condition associated with chronic liver disease other than HCV (such as but not limited to: hemochromatosis, autoimmune hepatitis,metabolic liver disease, alcoholic liver disease, toxin exposures)
* History of variceal bleeding, hepatic encephalopathy, or ascites requiring management with diuretics or paracentesis
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment
* Documented or suspected hepatocellular carcinoma (HCC)
* Positive for hepatitis B surface antigen (HBsAg)
* Positive for Human Immunodeficiency Virus-1 (HIV-1) and/or Human Immunodeficiency Virus-2 (HIV-2) antibodies
* Alanine transferase (transminase) (ALT) >5x upper limit of normal (ULN)
* Total Bilirubin ≥2 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) at 12 weeks post-treatment (SVR12) | 12 weeks post-treatment

SECONDARY OUTCOMES:
Proportion of subjects with HCV ribonucleic acid (RNA) < limit of quantification (LOQ) (detectable and undetectable) | Weeks 1, 2, 4, 6, 8, 10, 12,14, 16, 18, 20, 22 and 24 weeks of therapy; at end of treatment (EOT) (following 12 or 24 weeks of treatment, by Group); and Weeks 4, 12, 24, 36, and 48 weeks post-treatment
Proportion of subjects with HCV ribonucleic acid (RNA) undetectable | Weeks 1, 2, 4, 6, 8, 10, 12,14, 16, 18, 20, 22 and 24 weeks of therapy; at end of treatment (EOT) (following 12 or 24 weeks of treatment, by Group); and Weeks 4, 12, 24, 36, and 48 weeks post-treatment
Proportion of subjects who experience viral breakthrough | Formal analysis at SVR12, Week 48 of follow up period (or upon occurrence)
  viral breakthrough defined as:
  * Any increase in HCV RNA ≥ 1 log10 from nadir or
  * Any quantifiable HCV RNA ≥ 25 IU/mL (> LOQ) on or after Week 8
Proportion of subjects who experience viral relapse defined as confirmed quantifiable HCV RNA ≥ 25 IU/mL (>LOQ) in a subject with HCV RNA < LOQ or undetectable at End of treatment (EOT) | End of treatment (Maximum up to 24 Weeks)
Maximum observed plasma concentration (Cmax) of BMS-650032, BMS-790052, BMS 791325, and BMS-794712 | Day 1 and Day 14
Observed plasma concentration at 12 hours (C12) of BMS-650032, BMS-790052, BMS 791325, and BMS-794712 | Day 1 and Day 14
Observed plasma concentration at 24 hours (C24) of BMS-650032, BMS-790052, BMS 791325, and BMS-794712 | Day 1 and Day 14
Trough observed plasma concentration (Ctrough) of BMS-650032, BMS-790052, BMS 791325, and BMS-794712 | Day 1 and Day 14
Time of maximum observed plasma concentration (Tmax) of BMS-650032, BMS-790052, BMS 791325, and BMS-794712 | Day 1 and Day 14
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-650032, BMS-790052, BMS 791325, and BMS-794712 | Day 1 and Day 14
HCV genomic substitutions associated with exposure of BMS-650032, BMS-790052, and BMS-791325 | At the time of viral breakthrough or relapse
Frequency of deaths, serious adverse events (SAEs), discontinuations due to adverse events (AEs), severity Grade 3/4 AEs, and severity Grade 3/4 laboratory abnormalities | Formal analysis at week 48 of follow up period (or upon occurrence)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (26):
  - The Kirklin Clinic, Birmingham, Alabama
  - Southern California Research Center, Coronado, California
  - Peter J Ruane Md Inc, Los Angeles, California
  - Va Greater Los Angeles Healthcare System, Los Angeles, California
  - Research And Education, Inc., San Diego, California
  - Precision Research Institute, Llc, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - University Of Colorado Denver And Hospital, Aurora, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Orlando Immunology Center, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Atlanta Gastroenterology Associates, Llc, Atlanta, Georgia
  - Mercy Medical Center, Inc., Baltimore, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - Id Care, Hillsborough, New Jersey
  - Southwest Care Center, Santa Fe, New Mexico
  - James J Peters Vamc, The Bronx, New York
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Texas Clinical Research Institute, Arlington, Texas
  - Research Specialists Of Texas, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Metropolitan Research, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Dean Clinic, Madison, Wisconsin
- France (5):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Limoges
  - Local Institution, Marseille
  - Local Institution, Paris
- Fundacion De Investigacion De Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Everson GT, Sims KD, Thuluvath PJ, Lawitz E, Hassanein T, Rodriguez-Torres M, Desta T, Hawkins T, Levin JM, Hinestrosa F, Rustgi V, Schwartz H, Younossi Z, Webster L, Gitlin N, Eley T, Huang SP, McPhee F, Grasela DM, Gardiner DF. Daclatasvir + asunaprevir + beclabuvir +/- ribavirin for chronic HCV genotype 1-infected treatment-naive patients. Liver Int. 2016 Feb;36(2):189-97. doi: 10.1111/liv.12964. Epub 2015 Dec 6. PMID 26473667
- [Derived] Everson GT, Sims KD, Rodriguez-Torres M, Hezode C, Lawitz E, Bourliere M, Loustaud-Ratti V, Rustgi V, Schwartz H, Tatum H, Marcellin P, Pol S, Thuluvath PJ, Eley T, Wang X, Huang SP, McPhee F, Wind-Rotolo M, Chung E, Pasquinelli C, Grasela DM, Gardiner DF. Efficacy of an interferon- and ribavirin-free regimen of daclatasvir, asunaprevir, and BMS-791325 in treatment-naive patients with HCV genotype 1 infection. Gastroenterology. 2014 Feb;146(2):420-9. doi: 10.1053/j.gastro.2013.10.057. Epub 2013 Oct 30. PMID 24184132
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx